CLINICAL TRIAL: NCT02251444
Title: Emotionsregulation Und Bewältigungsverhalten in Zusammenhang Mit Ambulanter Rehabilitation Oder Physikalischer Therapie Bei Chronischem Rückenschmerz
Brief Title: Regulation of Emotions and Coping Behaviour in Patients With Chronic Recurrent Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment problems in the controle group
Sponsor: Karl Landsteiner Institute of Remobilization and Functional Health (Other)
Responsible Party: Principal Investigator, Michael Quittan, Prim. Univ. prof. Dr. Michael Quittan, Karl Landsteiner Institute of Remobilization and Functional Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rehabilitation program LBP
Record Dates: First submitted 2014-07-07; First posted 2014-09-29 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Physical Therapy Modalities

ARMS (2):
- outpatient rehabilitation program (Experimental): whole-body resistance training, psychological interventions, sessions for information related to ergonomics and healthy alimentation
  Interventions: Procedure: outpatient rehabilitation program
- physical therapy (Active Comparator): prescribed physical therapy
  Interventions: Procedure: physical therapy

INTERVENTIONS:
Procedure: outpatient rehabilitation program
  Arms: outpatient rehabilitation program
Procedure: physical therapy
  Arms: physical therapy

SUMMARY:
This study investigates effects of a multidisciplinary rehabilitation program or physical therapy in patients with chronic low back pain on emotion regulation and coping behaviour.

Hypothesis: Significant differences of negative emotions pre and post treatment and between groups after intervention.

Standardised questionnaires are used for investigation

DETAILED DESCRIPTION:
Emotionsregulations-Inventar ERI Emotion Regulation Questionnaire ERQ Positive and Negative Affect Schedule PANAS Brief Symptom Inventory BSI-18

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain > 3 months
* VAS >= 2
* understanding of german language

Exclusion Criteria:

* retired
* psychiatric disorders
* dementia
* sick headache
* chronic pain disease other than chronic low back pain
* patients with general contraindications of the therapy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Emotion regulation before and after treatment | 6-8 months
  Emotion regulation will be assessed with the questionnaire Emotionsregulations-Inventar ERI

SECONDARY OUTCOMES:
Isometric muscle strenght before and after treatment | 6-8 months
  The maximum voluntary isometric muscle strength of the lumbar extensor muscles will be assessed
Pain in the spine before and after treatment | 6-8 months
  Pain will be assessed with Visual Analogue Scale
Emotion regulation before and after treatment | 6-8 months
  Emotion regulation will be assessed with the Emotion Regulation Questionnaire ERQ

CONTACTS AND LOCATIONS:
Locations (1):
- Karl Landsteiern Institute of Remobilisation and Functional Health, Vienna, Vienna, Austria